CLINICAL TRIAL: NCT01132287
Title: An Evaluation of a Marketed Lubricated Eye Drop in Soft Contact Lens Wearers Who Experience Ocular Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SMA-09-50
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2012-01

CONDITIONS: Contact Lens Wear
Keywords: Contact lens wear; lubricant eye drops

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 FID 112903 (Experimental): FID 112903
  Interventions: Other: FID 112903
- No Intervention (No Intervention)

INTERVENTIONS:
Other: FID 112903 — lubricant eye drop FID 112903
  Other Names: Systane Ultra
  Arms: 1 FID 112903

SUMMARY:
Study to evaluate subjective comfort associated with the use of a marketed lubricant eye drop, by subjects reporting ocular dryness and wearing soft contact lenses on a daily disposable replacement schedule.

DETAILED DESCRIPTION:
The objective of this study is to evaluate subjective comfort associated with the use of a marketed lubricant eye drop, by subjects reporting ocular dryness and wearing soft contact lenses on a daily disposable replacement schedule.

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes

Exclusion Criteria:

* Topical ocular medication use Unstable or active ocular issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Subjective Comfort | 14 days

SECONDARY OUTCOMES:
Slit Lamp | 14 Days
Visual Acuity | 14 Days

REFERENCES:
- [Result] McDonald M, Schachet JL, Lievens CW, Kern JR. Systane(R) ultra lubricant eye drops for treatment of contact lens-related dryness. Eye Contact Lens. 2014 Mar;40(2):106-10. doi: 10.1097/ICL.0000000000000018. PMID 24552755